CLINICAL TRIAL: NCT00648869
Title: Open-label,Randomized, Crossover Study Comparing Metformin Gum and Immediate Release Tablet in Healthy Volunteers
Brief Title: Open-label Crossover Metformin Gum Versus Tablet in Healthy Volunteers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Drug was not sent
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Prof. Itamar Raz, Hadassah Medical Organization, Jerusalem, Israel
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: generex-HMO-CTIL
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2008-03

CONDITIONS: Healthy
Keywords: pharmaceutical preparations
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: metformin tablet, metformin gum — 500 mg, 250 mg

SUMMARY:
Single-dose, randomized, open-label, cross over study. The study will have an open-label, 3 period, 3 treatments, and randomized design.

Each volunteer will receive a Metformin gum 2x250mg, Metformin gum 1x250mg & Metformin tablet 500mg

ELIGIBILITY:
Inclusion Criteria:

* Men ranging in age from 18-40
* Good general health as determined by medical history, physical examination, ECG, Blood pressure, and clinical laboratory tests (hematology & clinical chemistry) obtained within 14 days prior to the start of the study.
* BMI >18&<30.
* Willing and able to abide by the dietary requirements of the study.
* Willing and able to give written informed consent in a manner approved by the Ethics Committee.

Exclusion Criteria:

* History of known or suspected clinically significant hypersensitivity to any drug.
* Any protocol-required laboratory test abnormality that is considered clinically significant.
* Mentally unstable or incompetent.
* Any illness during the week before.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-10 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
To determine the difference in the pharmacokinetic profile of metformin following administration of two formulations (gum and tablet). | 45 days

SECONDARY OUTCOMES:
To evaluate the effect on blood glucose levels as well as safety and tolerability of one time administration of the Metformin Gum and Metformin tablet. | 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Itamar Raz, MD, Principal Investigator — Hadassah Hebrew University Hospital
Locations (1):
- Diabetes Unit, Hadassah Hebew University Hospital, Jerusalem, Israel